CLINICAL TRIAL: NCT06104605
Title: Improving Access to Chiropractic Care for Low Back Pain in Underserved Primary Care Settings: A Protocol for a Pilot Study of a Multi-level Implementation Strategy
Brief Title: Improving Access to Chiropractic Care in Community Health Centers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-41930; K23AT010487 (NIH)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Lower Back Pain
Keywords: Chiropractic care; Primary care provider; Chiropractor referrals; Chronic pain; Non-pharmacologic treatment; Community health centers
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge design. 3 CHCs will be randomized to receive the intervention either first, second, or third two months apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation (Experimental): Implementation will be deployed at the CHC, PCP, and patient level.
  Interventions: Other: Institutional interventions; Other: PCPs interventions; Other: Patient interventions
- Standard of care (No Intervention): Usual patient care without deployment of intervention.

INTERVENTIONS:
Other: Institutional interventions — Intervention will include, but not be limited to, the following: adding a referral option to chiropractic care in the electronic health record (EHR), optimizing referral option, e.g., creating a list of preferred providers. Additional strategies may be added depending on community health center staff engagement prior to implementation.
  Arms: Implementation
Other: PCPs interventions — Two one-hour interactive grand rounds/lunch seminars that allow for inter-professional learning for PCPs with optional continuing education credits for PCPs.
  Short teaching cases involving clinical vignettes developed with local doctors of chiropractic (DCs), information about DCs (e.g., evidence-base for treatments), and logistics of the referral process (e.g., geographic location of community-based DCs who accept Medicaid) sent to participating providers unable to attend the seminars. Additional strategies may be added depending on primary care provider engagement prior to implementation.
  Arms: Implementation
Other: Patient interventions — Printed and electronic educational materials (e.g., brochures) written at a sixth grade reading level in English and Spanish that present chiropractic as a safe and effective evidence-based treatment for LBP. These materials will be written, reviewed, and revised by the researchers with CHC patient input. Additional strategies may be added depending on patient engagement prior to implementation.
  Arms: Implementation

SUMMARY:
The goal of this study is to evaluate the feasibility of new implementation strategies designed to increase the number of Primary Care Providers (PCPs) referrals to chiropractic care for lower back pain (LBP) in underserved populations. The investigators plan to pilot the strategies in three qualified community health centers (CHCs) and compare the number of LBP patients who receive referrals before and after implementation. The implementation strategies involve PCP, patient, and organizational interventions.

Patients presenting with LBP will be provided educational materials that focus on the safety and effectiveness of chiropractic care as an evidence-based treatment for LBP. Materials will be available in CHC common areas and may be sent to patients by their PCP via patient portal.

PCPs will participate in interactive lunch seminars to allow for inter-professional learning for PCPs. They will also participate in a survey regarding their attitudes and beliefs relating to chiropractic care. Currently, many PCPs cannot make chiropractic care referrals in the electronic health record (EHR). The investigators plan to add this option, or make it easier if the referral is already available.

This multi-level, multi-component approach will last two months, and will be rolled out sequentially in three clinics using a stepped-wedge design. The ordering of clinics will be random.

The primary outcome is the proportion of patients with LBP who received a referral to chiropractic care before and after the intervention. Secondary outcomes include referral to any non-pharmacologic treatment, use of imaging, and prescribed medications.

ELIGIBILITY:
Inclusion criteria for CHCs:

* Be a CHC in the Boston area with primary care
* Agree to participate in study

Inclusion criteria for PCPs:

* Work at a participating CHC
* Be an MD, doctor of osteopathy (DO), nurse practitioner (NP), or physician assistant (PA)

Inclusion criteria for patients with LBP:

* Has PCP at participating CHC
* Has LBP diagnosis
* Is 18 years of age or older

Exclusion criteria for CHCs:

* There are no exclusion criteria

Exclusion criteria for PCPs:

* There are no exclusion criteria

Exclusion criteria for patients with LBP:

* There are no exclusion criteria for adult patients with LBP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in PCP Chiropractor Referrals for LBP | During the fourteen month study period
  This outcome will be assessed by calculating the proportion of LBP patients receiving a chiropractic referral for the two timeframe periods will be calculated. The numerator will be those with a chiropractic referral, defined as those LBP patients who received a PCP referral in the EHR or documentation in the EHR of a visit with a chiropractor. The denominator will be the total number of unique LBP patients seen by a PCP with an LBP diagnosis in the EHR.

SECONDARY OUTCOMES:
Percentage of patient participants referred to physical therapy | 14 months
  Information for this outcome will be abstracted from the participants' medical records
Percentage of patient participants referred to acupuncture | 14 months
  Information for this outcome will be abstracted from the participants' medical records
Percentage of patient participants prescribed opioids | 14 months
  Information for this outcome will be abstracted from the participants' medical records
Percentage of patient participants referred to magnetic resonance imaging (MRI) | 14 months
  Information for this outcome will be abstracted from the participants' medical records
Percentage of patient participants that receive epidural injections | 14 months
  Information for this outcome will be abstracted from the participants' medical records

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Roseen, DC, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roseen EJ, Bussieres A, Reichman R, Bora C, Trieu J, Austad K, Williams C, Fischer RA, Parrilla D, Laird LD, LaValley M, Evans RL, Saper RB, Morone NE. A multi-level implementation strategy to increase adoption of chiropractic care for low back pain in primary care clinics: a randomized stepped-wedge pilot study protocol. Chiropr Man Therap. 2025 Feb 20;33(1):9. doi: 10.1186/s12998-024-00565-w. PMID 39979943